CLINICAL TRIAL: NCT06210685
Title: A Post-Market Study Evaluating Fluid Shunting Using the Automatic Continuous Effusion Management System (ACES™) in Patients With Symptomatic Aseptic Pleural Effusion
Brief Title: The ACES Study for Aseptic Pleural Effusion
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pleural Dynamics, Inc. (Industry)
Collaborators: Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL2301
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Pleural Effusion
Keywords: pleural effusion; malignant pleural effusion; IPC
MeSH Terms: conditions — Pleural Effusion; Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ACES Device (Experimental): Implantation of the ACES device for treatment of aseptic pleural effusion
  Interventions: Device: Automatic Continuous Effusion Shunt implantation

INTERVENTIONS:
Device: Automatic Continuous Effusion Shunt implantation — The catheter pump chamber is placed with part of the chamber between adjacent ribs and part of the chamber under the skin and external to the ribs. The pump chamber is used to transfer pleural fluid into the peritoneal cavity.
  Other Names: ACES Catheter

SUMMARY:
The study will enroll recurrent aseptic pleural effusion patients who are designated by their physician as needing treatment to control the fluid. Baseline assessment will include a history and physical, chest imaging and quality of life questionnaires.

After ACES implantation, patients will remain under hospital care for general observation as per standard-of-care before being discharged home with access to electronic diaries for tracking pain and dyspnea.

DETAILED DESCRIPTION:
Pleural Dynamics is the first company to provide a fully implantable automatic effusion shunt that is powered by normal breathing and is designed for continuous symptom relief, and does not require an extended hospital stay, a catheter external to the chest, or expensive drainage canisters."

The current standard of care, pleurodesis, is often painful, requires an extended hospital stay, and is often unsuccessful requiring additional procedures to manage the effusion1. While an alternate approach-indwelling pleural catheters-exists, it requires that the patient have a portion of the catheter to be external to the chest and requires frequent drainage into proprietary external canisters to relieve symptoms. Pleural Dynamics' patented ACES™ System addresses these shortcomings with its' one-piece, fully implanted system that can be placed during a short hospital stay. This technology is designed to use normal breathing motion to automatically pump pleural effusion fluid out of the chest to the abdomen for reabsorption by the body eliminating the need for an external catheter and frequent drainage, providing ongoing symptom relief.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent pleural effusion after thoracentesis for which the physician has determined that a catheter implantation is indicated.
2. Symptoms of PE such as shortness of breath, cough, or chest fullness/chest discomfort based on patient report to physician.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
4. Patient is willing and able to meet all study requirements, including follow-up visits and receiving study related telephone calls.

Exclusion Criteria:

1. Recurrent pleural effusion after thoracentesis for which the physician has determined that a catheter implantation is indicated.
2. Symptoms of PE such as shortness of breath, cough, or chest fullness/chest discomfort based on patient report to physician.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
4. Patient is willing and able to meet all study requirements, including follow-up visits and receiving study related telephone calls.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | 30 days
  Percentage change in pleural effusion volume via chest CT from baseline

SECONDARY OUTCOMES:
Adverse Events | 30 and 60 days
  Rate of Adverse Events (serious and non-serious) including hospitalizations/visits
Pleurodesis | 30 and 60 days
  Rate of Pleurodesis
VAS Breathlessness Score | 30 and 60 days
  Change in VAS Breathlessness Score

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Moldanado, MD, MSc, Principal Investigator — Vanderbilt University
Locations (4):
- United States (4):
  - Memorial Healthcare System, Hollywood, Florida
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - University of North Carolina Pulmonary and Critical Care Medicine, Chapel Hill, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No